CLINICAL TRIAL: NCT01491100
Title: Study Assessing Cognitive Performance Plus Physical Activity in Patients With Relapsing-Remitting MS Under Treatment With Betaferon®
Brief Title: Noninterventional Study Assessing Cognitive Function and Physical Activity in People With Multiple Sclerosis
Acronym: CogniPlus
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16036; BF1101 (Other: company internal)
Record Dates: First submitted 2011-12-12; First posted 2011-12-13 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
Keywords: Cognition; Physical Activity; Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Patients treated with regular dose subcutaneously administered, according to the label and to clinical routine practice.

SUMMARY:
Study assessing cognitive function and physical activity in people with relapsing remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Relapsing Remitting Multiple Sclerosis (RRMS), and treated with Betaferon, with the decision for treatment made at the discretion of the attending physician, documented with a prescription of Betaferon by the physician
* EDSS 0 - 6
* Written informed consent

Exclusion Criteria:

* Patients who do not meet the local indication criteria for Betaferon treatment.
* Contraindications listed in the local SmPCs have to be considered.
* Patients with a history of severe head trauma.
* Patients with alcohol and/or drug abuse.
* Patients with mental retardation.
* Patients with learning disability.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 1085 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Cognitive performance as measured by SDMT (Symbol Digit Modalities Test) | 24 months
Physical activity as measured by the Baecke questionnaire | 24 months

SECONDARY OUTCOMES:
Disability as measured by EDSS (Expanded Disability Status Scale) | 24 months
Fatigue as measured by FSMC (Fatigue Scale for Motor and Cognitive Functions) | 24 months
Depression as measured by the CES-D (Center for Epidemiologic Studies Depression) | 24 months
Quality of life as measured by the SF-12 (Mental and physical health-scale measure of quality of life) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (17):
- Multiple Locations, Albania
- Multiple Locations, Algeria
- Multiple Locations, Argentina
- Multiple Locations, Belgium
- Multiple Locations, Czechia
- Multiple Locations, Egypt
- Multiple Locations, France
- Multiple Locations, Germany
- Multiple Locations, Greece
- Multiple Locations, Hungary
- Multiple Locations, Israel
- Multiple Locations, Kazakhstan
- Multiple Locations, Netherlands
- Multiple Locations, Portugal
- Multiple Locations, Saudi Arabia
- Multiple Locations, Tunisia
- Multiple Locations, Turkey (Türkiye)